CLINICAL TRIAL: NCT02692339
Title: Prospective Observational Study Evaluating the Safety of Lenalidomide/Dexamethasone Treatment in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Safety Study of Lenalidomide/Dexamethasone to Treat Patients With Relapsed or Refractory Multiple Myeloma
Acronym: PrObe-L
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-5013-MM-028
Record Dates: First submitted 2016-02-22; First posted 2016-02-26 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Multiple Myeloma; Refractory Multiple Myeloma; Lenalidomide; Dexamethasone; Observational Study; Safety of Len/Dex
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lenalidomide/Dexamethasone: Standard of Care doses for relapsed/refractory multiple myeloma
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — Standard of Care doses for relapsed/refractory multiple myeloma: 25 mg/day lenalidomide 21 of 28 days cycle
  Other Names: Revlimid
Drug: Dexamethasone — Standard of Care doses for relapsed/refractory multiple myeloma: dexamethasone 40 mg/day at day 1,8,15,22 at 28 days cycle
  Other Names: Decadron

SUMMARY:
Multicentre, prospective, observational, open-label, single arm, post-marketing study intended to record Lenalidomide/Dexamethasone treatment data from patients with relapsed/refractory Multiple Myeloma (rrMM) treated under the settings defined by the standard clinical practice and approved Summary of Product Characteristics (SmPC).

DETAILED DESCRIPTION:
This study aims to assess the real-life safety of Lenalidomide/Dexamethasone (Len/Dex) in patients with (Relapsed or Refractory Multiple Myeloma (rrMM), by evaluation of adverse events of special interest (infections, gastrointestinal events, thrombocytopenia, neutropenia, febrile neutropenia, and thromboembolism). In addition, due to the scarce information regarding the impact of frailty in Len/Dex treatment in rrMM, this study will prospectively assess Len/Dex safety and effectiveness by patient frailty groups.

The following study assessments will be performed:

* Recruitment: patients will be recruited within 15 days after the start of Len/Dex (from day 1 to day 15). In case patients are not recruited at the day of Len/Dex start (day 1), baseline information respective to this day will be collected retrospectively.
* Treatment period: during this period, the following assessments will be carried out:

  * Every 30 days (± 5 days) for adverse events, changes in concomitant medication and change in Len/Dex dose.
  * Every 90 days (± 15 days) for the remaining information to be collected in the treatment period
* Assessment at the end of Len/Dex treatment (until 5 days after end of treatment).

Follow-up assessment 90 days (± 15 days) after the end of Len/Dex treatment.

No visits were predefined for this study. Study data is planned to be collected when the patient goes to the study site for a clinical routine visit. No assessments will be imposed for the purposes of this study. If the patient goes to the clinical routine visit at a date out of the time intervals predicted above, no information will be collected. Information will be collected in the context of routine clinical practice.

The patient will be followed until the end of Len/Dex treatment, death or discontinuation for any reason for a maximum period of 36 months, Patients within treatment after this maximum period will stop being followed in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or higher.
2. Patients who have voluntarily given written informed consent to participate in the study and have their data retrieved for the purposes of the study
3. Patients diagnosed with 1st or 2nd relapsed or refractory multiple myeloma and indicated for 2nd or 3rd line Len/Dex treatment, according with the SmPC (patients who have received at least one prior therapy) -

Exclusion Criteria:

1. Pregnant or lactating patients
2. Female patients of childbearing potential unable or unwilling to use effective contraceptive methods, as stated in the summary of product characteristics:

   * Implant.
   * Levonorgestrel-releasing intrauterine system.
   * Medroxyprogesterone acetate depot.
   * Tubal sterilisation.
   * Sexual intercourse with a vasectomised male partner only; vasectomy must be confirmed by two negative semen analyses.

   Ovulation inhibitory progesterone-only pills (i.e. desogestrel).

   - Male patients unable to follow or comply with the required contraceptive measures stated in the SmPC (use of condom if engaged in sexual activity with a pregnant woman or a woman of childbearing potential not using effective contraception [even if the man has had a vasectomy], during treatment and for 1 week after dose interruptions and/or cessation of treatment)
3. Hypersensitivity to the active substance or any of the excipients
4. Patients participating in a clinical trial -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relapsed and/or Refractory multiple myeloma patient population
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events of special interest during Len/Dex therapy | Up to approximately 72 months
  Adverse event (AE): Any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment, i.e. any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product whether or not considered related to the medicinal product. Progression of the underlying disease of multiple myeloma is not considered an AE and should not be reported as an AE

SECONDARY OUTCOMES:
Incidence (number) of thromboembolism | Up to approximately 72 months
  Identification of the incidence of deep venous thrombosis and pulmonary embolism) during Lenalidomide and Dexamethasone study drug treatment.
Duration of Len/Dex treatment over the course of the study | Up to approximately 72 months
  Defined as the time between the start of Len/Dex treatment until discontinuation or death (whichever occurs first)
Number of patients with good and poor compliance to lenalidomide and dexamethasone | Up to approximately 72 months
  Compliance will be measured by the capsule/tablet count, after the end of study treatment
Type and frequency of prophylaxis treatment for prevention of thromboembolism | Up to 36 months
  Type and frequency of prophylaxis treatment for prevention of thromboembolism during Lenalidomide/Dexamethasone study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Boaventura, MD, Study Director — Celgene
Locations (12):
- Portugal (12):
  - Hospital Garcia Orta, E.P.E., Almada
  - Hospital Professor Doutor Fernando Fonseca, E.P.E., Amadora
  - Hospital Central de Faro, Faro
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, EPE, Lisbon
  - Centro Hospitalar Lisboa Central, EPE - Hospital de Sto. Ant. Capuchos, Lisbon
  - Fundação Champalimaud, Lisbon
  - Centro Hospitalar Lisboa Norte, EPE - Hospital Santa Maria, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar de São João, EPE - Hospital de São João, Porto
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
  - Hospital de São Teotónio, E.P.E., Viseu